CLINICAL TRIAL: NCT03196830
Title: Safety and Efficacy of Chimeric Antigen Receptor T Cell (CAR-T) Treating Relaspe/Refractory CD19/CD20/CD22/CD30 Postive Non-Hodgkin Lymphoma
Brief Title: CAR-T for R/R B-NHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ5601
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; CAR - T CD19/CD20/CD22/CD30
Keywords: Relapse/refractory non-Hodgkin lymphoma; CAR - T CD19/CD20/CD22/CD30
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): the group of patients who received CAR-T treatment
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — For eligible patients, CAR-T cells targeted to patients' tumor cell antigen will be infused after 48 hours later of chemotherapy

SUMMARY:
This study is a single arm study to investigate the efficacy and safety of CAR-T targeted CD19/CD20/CD22/CD30 in relapse and refractory non-Hodgkin lymphoma patients. Ten patients will recruieted, admitted in hospital for 1 month for the CAR-T treatment and follow-up for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological detection confirmed CD19/CD20/CD22/CD30 postive non-Hodgkin lymphoma
* Recieved more than 2 lines of chemotherapy
* With contraindications of hematopoietic stem cell transplantation or relapse after hematopoietic stem cell transplantation
* Expected survival more than 3 months
* Karmofsky performance score ≤ 60, and ECOG ≥ 2.
* Enough organ function: EF≥50%; normal ECG; CCR≥40ml/min; ALT and AST ≤ 3 × upper limitation of normal, T-BIL ≤ 2.0mg/dl; PT and APTT < 2 × upper limitation of normal; SpO2 > 92%
* CBC results: Hb ≥ 80g/L, ANC > 1 × 10E9/L, Plt ≥ 50 × 10E9/L
* Results of pregnant test should be negative, and agree to conception control during treatment and 1 year after CAR-T infusion
* With measurable disease
* Written informed consent could be acquired

Exclusion Criteria:

* Received immunol suppression treatment or steroids in recent 1 week before recruitment
* Uncontrolled infection
* HIV positive patients
* Active HBV or HCV infection
* Women in pregnancy and lactation
* Refuse to conception control during treatment and 1 year after CAR-T infusion
* Uncured malignancies other than non-Hodgkin lymphoma
* Have participated similar trial for treating relapse/refractory non-Hodgkin lymphoma
* Inheritated immune deficiancy
* Severe heart disease

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | One months after CAR-T cells were infused
  Rate of complete remission and patial remission

SECONDARY OUTCOMES:
Adverse toxicity | Day 0, day 4, week 1, week 3, week 4, month 2, month 24 after CAR-T cells were infused
  Accordingto CTCAE 4.0 criteria
CAR-T cell survival | every week in first 4 weeks after CAR-T cells infusion, then every 3 months for 2 years, then every 6 months for next 2 years
  the survival of CAR-T cells detected in patients' peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou J, Zhang Y, Shan M, Zong X, Geng H, Li J, Chen G, Yu L, Xu Y, Li C, Wu D. Cytopenia after chimeric antigen receptor T cell immunotherapy in relapsed or refractory lymphoma. Front Immunol. 2022 Sep 5;13:997589. doi: 10.3389/fimmu.2022.997589. eCollection 2022. PMID 36131934
- [Derived] Sang W, Wang X, Geng H, Li T, Li D, Zhang B, Zhou Y, Song X, Sun C, Yan D, Li D, Li Z, Li C, Xu K. Anti-PD-1 Therapy Enhances the Efficacy of CD30-Directed Chimeric Antigen Receptor T Cell Therapy in Patients With Relapsed/Refractory CD30+ Lymphoma. Front Immunol. 2022 Apr 1;13:858021. doi: 10.3389/fimmu.2022.858021. eCollection 2022. PMID 35432352
- [Derived] Zhang Y, Li J, Lou X, Chen X, Yu Z, Kang L, Chen J, Zhou J, Zong X, Yang Z, Li M, Xu N, Jia S, Geng H, Chen G, Dai H, Tang X, Yu L, Wu D, Li C. A Prospective Investigation of Bispecific CD19/22 CAR T Cell Therapy in Patients With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma. Front Oncol. 2021 May 25;11:664421. doi: 10.3389/fonc.2021.664421. eCollection 2021. PMID 34113569
- [Derived] Li C, Zhang Y, Zhang C, Chen J, Lou X, Chen X, Kang L, Xu N, Li M, Tan J, Sun X, Zhou J, Yang Z, Zong X, Wang P, Xu T, Qu C, Huang H, Jin Z, Yu L, Wu D. Comparation of CART19 and autologous stem-cell transplantation for refractory/relapsed non-Hodgkin's lymphoma. JCI Insight. 2019 Jul 23;5(17):e130195. doi: 10.1172/jci.insight.130195. PMID 31335321
- [Derived] Qu C, Ping N, Kang L, Liu H, Qin S, Wu Q, Chen X, Zhou M, Xia F, Ye A, Kong D, Li C, Yu L, Wu D, Jin Z. Radiation Priming Chimeric Antigen Receptor T-Cell Therapy in Relapsed/Refractory Diffuse Large B-Cell Lymphoma With High Tumor Burden. J Immunother. 2020 Jan;43(1):32-37. doi: 10.1097/CJI.0000000000000284. PMID 31219975